CLINICAL TRIAL: NCT01315262
Title: On Demand Versus Daily Sildenafil for Patients Undergoing Bilateral Nerve Sparing Radical Prostatectomy: a Randomized, Open Label, Parallel Group Trial
Brief Title: On Demand Versus Daily Sildenafil for Patients Undergoing Radical Prostatectomy
Acronym: URO2010
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: francesco montorsi, Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR Urology
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-02

CONDITIONS: Erectile Dysfunction
Keywords: Sildenafil 100; restoring erectile function after radical prostatectomy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viagra 100 mg daily (Active Comparator)
  Interventions: Drug: Sildenafil
- Viagra 100mg on demand (Active Comparator)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 1:1 Viagra 100 mg daily (taken either at bedtime - if sexual intercourse is not expected - or 1 hour prior to sexual intercourse, no more than one 100 mg dose of sildenafil per day) vs. Viagra 100mg OD (i.e. one hour prior to sexual intercourse)

SUMMARY:
Viagra (Sildenafil citrate) is an orally active selective inhibitor of cyclic guanosine monophosphate (cGMP)-specific phosphodiesterase type 5 (PDE5) which is used for the treatment of erectile dysfunction (ED). Objectives:

* To test the efficacy of Viagra 100mg on demand vs. Viagra 100mg daily (taken either at bedtime or 1 hour prior to sexual intercourse) in restoring erectile function following radical prostatectomy.
* To test the safety and tolerability of Viagra 100 mg on demand vs. Viagra 100 mg daily after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have given written informed consent to participate in the study.
2. Men aged 18-65 years old.
3. Weight range 50-100 Kg.
4. Subjects must be in a stable relationship with the same partner for at least 6 months and willing to attempt sexual intercourse.
5. Normal pre-operative erectile function (defined as IIEF-EF ≥ 26) without the use of therapy or devices for the improvement of erections.
6. Prostatic Specific Antigen (PSA) lower than 10 ng/ml.
7. Clinical prostate cancer stage T1c or T2.
8. Biopsy Gleason sum < 8.
9. Able to read, understand and provide signed informed consent.

   Intra-operative inclusion criteria:
10. Bilateral nerve sparing radical prostatectomy (both open and robotic assisted radical prostatectomy are accepted) as defined by the surgeon.

    Post-operative inclusion criteria:
11. Histologically-confirmed, organ-confined prostate cancer disease (defined as, Gleason 6 or 7 and, pathological stage T2 or T3a R0 N0).

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Subjects in whom sexual activity is inadvisable in the opinion of the investigator such as significant cardiovascular disease in the last 6 months; including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischemic attack (TIA), symptomatic or clinically significant cardiac arrhythmias including atrial fibrillation.
2. Subjects who have a medical history of major hematological, renal, vascular or hepatic abnormalities, those with psychological or social circumstances that would impair their ability to participate reliably in the study, or those who may increase the risk to themselves or others by participating in the study.
3. Subjects who have a medical history of diabetes.
4. Subjects who developed a postoperative complication, namely reoperation for hemorrhage, a documented urinary fistula or the indwelling of catheter for 3 or more weeks.
5. Subjects treated with neo-adjuvant radiotherapy or hormonotherapy.
6. Subjects who have received or are receiving any PDE5 inhibitors.
7. Subjects with known hypersensitivity to Viagra or any component of the study medication.
8. Subjects with resting sitting hypotension (BP < 90/50 mmHg), hypertension (BP > 170/110 mmHg) or orthostatic hypotension.
9. Subjects with severe hepatic; cirrhosis or ALT (Alanine aminotransferase) 2x upper limit of normal) and renal impairment (creatinine clearance 30mL/min) or known history of hereditary degenerative retinal disorders such as retinitis pigmentosa.
10. Subjects who, for medical reasons and/or in the opinion of the investigator, require starting dose of 25mg of Viagra.
11. Subjects who are currently taking or are likely to be treated with nitrates or nitric oxide donors in any form (oral, sublingual, buccal, transdermal, inhalational or as aerosols) on either regular or intermittent basis.
12. Subjects who are receiving concomitant treatment or who during the study are likely to start the treatment with potent CYP3A4 and CYP2C9 inhibitors (e.g. protease inhibitors ritonavir and saquinavir, ketoconazole, itraconazole, Miconazole, nefazadone, claritromycin, troleandomycin erythromycin and cimetidine).
13. Subjects who are currently using any commercially available treatments or non-commercial herbal preparations for erectile dysfunction, e.g. IC injections, vacuum devices, or testosterone patches. Such treatments/devices must not be used at any time during the study.
14. Subjects who have received any investigational drug within the six weeks prior to screening or who are taking any other investigational drug concomitantly.
15. previous prostate surgery or previous hormonal treatment.
16. Subjects at increased risk of priapism e.g. sickle cell disease, multiple myeloma, or with anatomical deformation of the penis (such as angulation, cavernosal fibrosis or Peyronie's disease) and myeloproliferative disorders (e.g. myeloid leukemia, polycythemia, thrombocytopenia).
17. Subjects with other forms of sexual dysfunction (e.g. retrograde ejaculation, unejaculation, painful ejaculation, premature ejaculation, hypoactive sexual desire and inhibited or absent orgasm).
18. Subjects who, in the opinion of the investigator, abuse alcohol or drugs.
19. Subjects who, in the opinion of the investigator, are not likely to complete the event logs and follow study instructions.
20. Subjects who, in the opinion of the investigator, are not likely to complete the study for whatever reason.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an Erectile Function domain score of International Index of Erectile Function ( IIEF) => 22 at the end of the wash-out period (44 wks after surgery) | 44 wks after surgery

SECONDARY OUTCOMES:
Proportion of patients with an Erectile Function domain score of IIEF => 22 at the end of the study (52 wks after surgery) | 52 wks after surgery
IIEF - Domain Scores for: Erection Hardness Score (1-4) Intercourse success rates defined by the Sexual Encounter Profile (SEP) questionnaire (questions 2 and 3) Safety Endpoints: Adverse event summarized Global assessment questions | 3-6-9-12 months
  Responses to IIEF - Domain Scores for:
  * Erectile Function
  * Orgasmic Function
  * Sexual Desire
  * Intercourse Satisfaction
  * Overall Satisfaction c. Erection Hardness Score
  * Intercourse success rates defined by the SEP questionnaire (questions 2 and 3)
  * Safety Endpoints: Adverse event data will be summarized
  * Global assessment questions:

CONTACTS AND LOCATIONS:
Overall Officials: francesco montorsi, MD, Principal Investigator — Vita-Salute San Raffaele Hospital
Locations (1):
- Vita-Salute San Raffaele, Milan, Italy